CLINICAL TRIAL: NCT00059241
Title: Reach For Health--Middle Childhood Risk Prevention Study
Brief Title: The "Reach For Health" Program: Delaying Sexual Activity in Children
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5R01HD39537-2; 5R01HD039537 (NIH)
Record Dates: First submitted 2003-04-22; First posted 2003-04-23 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-04

CONDITIONS: Sex Behavior; Child Behavior
Keywords: Early sexual initiation; Prevention of early sexual activity; Middle childhood
MeSH Terms: conditions — Sexual Behavior; Child Behavior

INTERVENTIONS:
Behavioral: Parent-child communication education
Behavioral: Service learning
Behavioral: Classroom health curriculum

SUMMARY:
Working with multiple schools in Brooklyn, NY, this study will develop and evaluate school- and community-based strategies designed to reduce early sexual activity and risky sexual behavior in middle school-aged children. These strategies will focus on parent education, classroom health curriculum, and learning through participation in community service.

DETAILED DESCRIPTION:
Given the early age of sexual initiation among urban minority youth, interventions aimed at reducing sexual initiation and risky sexual behavior related to HIV and other sexually transmitted infections (STIs) should begin prior to entry into middle school. These interventions should support both students and their parents through the transition to early adolescence. In collaboration with the New York City Public Schools, this study is designed to evaluate strategies to prevent early sexual initiation and its precursors among academically at-risk urban minority boys and girls.

This study will answer two questions: 1) do factors that predict sexual risk taking and its precursors in young adolescence operate similarly in middle childhood; and 2) can interventions shown to be effective in early adolescence be developmentally adapted for middle childhood to delay sexual initiation and its precursors? The study will evaluate the impact of the intervention on mechanisms hypothesized to reduce sexual risk taking and its precursors, including the personal resiliency and social competencies of youth. The study will also collect data on the costs and process of implementation to inform subsequent dissemination.

Participants in this study will be fifth and sixth grade children enrolled in participating public schools in Brooklyn, NY. Participating school communities will be predominantly African American and Latino. In the fall of their fifth and sixth grade years, students and their families are assigned at random to participate in either a parent education group or in a control group. The parent education program, "Saving Sex for Later," focuses on the transition from middle childhood to early adolescence, the pressures to engage in risk behaviors (including early sexual initiation and related risks), and peer and parental influences on youth attitudes and behaviors. Those in the control condition receive a classroom health curriculum. In addition, a subgroup in each grade level is assigned to participate in service learning, an educational method in which personal and community values are taught through experience in structured service activities.

Youth will be followed for 12 to 18 months. Surveys will be conducted in the fall of the fifth and sixth grade years and again at a 3-month post intervention follow-up. These surveys will measure youth attitudes and behaviors, including precursors to early sexual initiation and related risk behaviors. Surveys of parents' attitudes and behaviors will also be conducted to supplement information from youth. To assist in interpreting results of the surveys, in-depth qualitative interviews will be conducted with a subgroup of fifth grade youth; these youth will be resurveyed prior to entry into seventh grade.

ELIGIBILITY:
Inclusion Criteria

* Youth attending NYC schools implementing "Reach for Health" program components and their parents
* Enrolled in general education classes
* Ability to complete survey assessments in English

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200
Dates: Start 2000-07

CONTACTS AND LOCATIONS:
Overall Officials: Lydia O'Donnell, Ed.D., Principal Investigator — Education Development Center, Inc.
Locations (1):
- Education Development Center, Inc., Newton, Massachusetts, United States